CLINICAL TRIAL: NCT00541164
Title: Effects of Coenzyme Q10 (CoQ10) on Subjects With Charcot-Marie-Tooth Disease (CMT):A Double Blind, Randomized, Controlled Trial With an Open Label Follow-up Study
Brief Title: Effects of Coenzyme Q10 on Charcot-Marie-Tooth Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 05-19
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2010-06

CONDITIONS: Charcot Marie Tooth Disease
Keywords: CMT; Charcot-Marie Tooth; CoQ10; Coenzyme Q10
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 300 mg CoQ10 chewable wafer twice a day
  Interventions: Drug: Coenzyme Q10
- 2 (Placebo Comparator): Chewable placebo wafer twice a day for 24 weeks with crossover to 300mg CoQ10 twice a day for weeks 24-48.
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Drug: Coenzyme Q10 — 300 mg CoQ10 twice a day for 48 weeks
  Other Names: CoQ10; Ubiquinone
  Arms: 1
Dietary Supplement: Coenzyme Q10 — 300mg CoQ10 twice a day for 24 weeks beginning at week 24 of the study
  Other Names: CoQ10; Ubiquinone
  Arms: 2

SUMMARY:
The object of this research is to test the effectiveness of Coenzyme Q10 (CoQ10) on symptoms of weakness, fatigue, and pain in persons with Charcot-Marie-Tooth disease (CMT).In this study we also intend to examine the impact of daily supplementation on overall quality of life.We are also interested in identifying any differences in serum ratios of CoQ10 in the oxidized and reduced forms.

DETAILED DESCRIPTION:
CoQ10 is an integral part of the electron transport chain in the mitochondria, or the energy production centers of cells. Within recent years, there has been expanding interest in the potential benefits of CoQ10 supplementation on a variety of neuromuscular diseases, some of which involve mitochondrial dysfunction, such as CMT. Daily supplementation may have cytoprotective and neuroprotective properties, which may improve symptoms of weakness, fatigue, and pain, as well as increase quality of life (QOL) among persons with CMT.

With regards to within group comparisons we hypothesize that daily supplementation of CoQ10 taken as a 300 milligram wafer twice a day for 3 months will produce a statistically significant reduction in weakness, fatigue, and pain, along with a significant improvement in QOL as indicated from scores in both standardized physiological and scale measures.

The addition of serum level analysis will help to contextualize clinical results. We hypothesize the ratios of the oxidized and reduced forms of CoQ10 will be modified upon supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of CMT, confirmed by review of medical records by the study physician
* Subjects can be of either gender
* Subjects must be between the ages of 18 and 75
* Subjects must be able to complete all assessments at the designated time intervals
* Subjects must review and sign the informed consent statement according to Conemaugh Memorial Medical Center's (CMMC) Institutional Review Board (IRB) guidelines
* Subjects must receive approval from their primary care physician (PCP) to enroll in the study
* Regarding weakness, fatigue, and pain, subjects must experience at least two of the three symptoms on most days over the past month
* Regarding weakness, fatigue, and pain, subjects must report experiencing maximum levels of >/= 3.0 centimeters (cm) on the 10 cm visual analog scale (VAS) for any two of the three symptoms over the past month
* Female subjects must be willing to practice stable birth control during involvement in the study
* Subjects must agree to be randomized

Exclusion Criteria:

* Subjects having another general medical condition, which might confound the assessment of weakness, fatigue, and pain due to CMT
* Subjects taking warfarin or Coumadin
* Subjects who are pregnant, verified by a urine pregnancy test*
* Subjects having a cognitive impairment scoring < 20 on the Mini-Mental State Exam
* Subjects who are currently using CoQ10 supplementation or have used it in the past 6 months
* Subjects with a history of chronic liver disease or other condition causing malabsorption
* Drug intake that could modify lipid absorption (such as statins)
* Subjects who consume >3 alcoholic drinks per day on more than one occasion per month
* Subjects with abnormal liver function tests as defined through a Hepatic -Function Panel or a Liver Function Panel

  * Women of childbearing age who have had at least one menstrual cycle within the past 12 months and who have not undergone a sterilization procedure will undergo a urine pregnancy test at visits 1-10 regardless of group assignment in order to maintain the single blind. The urine samples will be processed at CMMC's lab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Changes in weakness, fatigue and pain in persons with Charcot-Marie-Tooth disease after supplementation with 600 mgs a day of Coenzyme Q10. | 60 weeks

SECONDARY OUTCOMES:
Improvements in quality of life in subjects with CMT before and after CoQ10 supplementation. | 60 weeks
Measure blood serum levels of the oxidized and reduced forms of CoQ10. | 60 weeks
Measure liver function tests | visits 1, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Plank, MD, Principal Investigator — John P. Murtha Neuroscience and Pain Institute
Locations (1):
- John P Murtha Neuroscience and Pain Institute, Johnstown, Pennsylvania, United States

REFERENCES:
- [Background] Hendler SS, Rorvik D, eds. PDR for Nutritional Supplements. Montvale, NJ: Thomson PDR; 2001:105-106.
- [Background] Chaudhuri A, Behan PO. Fatigue in neurological disorders. Lancet. 2004 Mar 20;363(9413):978-88. doi: 10.1016/S0140-6736(04)15794-2. PMID 15043967
- [Background] Beal MF. Coenzyme Q10 as a possible treatment for neurodegenerative diseases. Free Radic Res. 2002 Apr;36(4):455-60. doi: 10.1080/10715760290021315. PMID 12069110
- [Background] Shults CW. Coenzyme Q10 in neurodegenerative diseases. Curr Med Chem. 2003 Oct;10(19):1917-21. doi: 10.2174/0929867033456882. PMID 12871093
- [Background] Bhagavan HN, Chopra RK. Coenzyme Q10: absorption, tissue uptake, metabolism and pharmacokinetics. Free Radic Res. 2006 May;40(5):445-53. doi: 10.1080/10715760600617843. PMID 16551570
- [Background] Shults CW, Oakes D, Kieburtz K, Beal MF, Haas R, Plumb S, Juncos JL, Nutt J, Shoulson I, Carter J, Kompoliti K, Perlmutter JS, Reich S, Stern M, Watts RL, Kurlan R, Molho E, Harrison M, Lew M; Parkinson Study Group. Effects of coenzyme Q10 in early Parkinson disease: evidence of slowing of the functional decline. Arch Neurol. 2002 Oct;59(10):1541-50. doi: 10.1001/archneur.59.10.1541. PMID 12374491
- [Background] Huntington Study Group. A randomized, placebo-controlled trial of coenzyme Q10 and remacemide in Huntington's disease. Neurology. 2001 Aug 14;57(3):397-404. doi: 10.1212/wnl.57.3.397. PMID 11502903
- [Background] Jones K, Hughes K, Mischley L, McKenna DJ. Coenzyme Q-10: efficacy, safety, and use. Altern Ther Health Med. 2002 May-Jun;8(3):42-55; quiz 56, 138. No abstract available. PMID 12017500
- [Background] Lagendijk J, Ubbink JB, Vermaak WJ. Measurement of the ratio between the reduced and oxidized forms of coenzyme Q10 in human plasma as a possible marker of oxidative stress. J Lipid Res. 1996 Jan;37(1):67-75. PMID 8820103